CLINICAL TRIAL: NCT01743222
Title: Cx621-0101 Phase I Clinical Trial in Healthy Volunteers to Evaluate the Feasibility and Safety of the Intralymphatic Administration Technique of Expanded Allogeneic Adipose-derived Stem Cells (eASCs)
Brief Title: Intralymphatic eASC Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Cx621-0101
Record Dates: First submitted 2012-08-24; First posted 2012-12-06 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Localized Adverse Reaction to Administration of Drug
MeSH Terms: interventions — hypothermosol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- eASC (Experimental): eASC
  * First cohort (3 volunteers, first volunteer is not randomized to detect any acute reaction): injection of 2.5 millions of eASCs suspended in 0.25 ml of HTS per lymph node, total dose 5 millions of cells.
  * Second cohort (3 volunteers, first volunteer is not randomized to detect any acute reaction): injection of 5 millions of eASCs suspended in 0.5 ml of HTS per lymph node, total dose 10 millions of cells.
  Interventions: Genetic: eASC
- Placebo (Placebo Comparator): * First cohort (2 volunteers): injection of 0.25 ml of Hypo Thermosol (HTS) per lymph node
  * Second cohort (2 volunteers): injection of 0.5 ml of Hypo Thermosol (HTS) per lymph node
  Interventions: Drug: Placebo

INTERVENTIONS:
Genetic: eASC — * First cohort: Intra lymph node injection of 2.5 millions of eASCs suspended in 0.5 ml of HypoThermosol per lymph node, total dose 5 millions of cells.
  * Second cohort: Intra lymph node injection of 5 millions of eASCs suspended in 0.25 ml of HypoThermosol per lymph node, total dose 10 millions of cells.
  Other Names: Allogenic Stem Cells
  Arms: eASC
Drug: Placebo — * First cohort (2 volunteers): injection of 0.25 ml of HypoThermosol (HTS) per lymph node
  * Second cohort (2 volunteers): injection of 0.5 ml of HypoThermosol (HTS) per lymph node
  Other Names: HypoThermosol HTS
  Arms: Placebo

SUMMARY:
The objective is to determine the safety, tolerability and feasibility of the inguinal intralymphatic administration of expanded allogeneic adipose-derived stem cells (eASCs)

DETAILED DESCRIPTION:
Phase I, unicentric, single blind, clinical trial with healthy volunteers to determine the feasibility of a new administration technique.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 both included
* Inform Consent Form signed
* Body Mass Index (BMI) between 19 and 29 kg/m2
* Presence of, at least, one lymph node of 1cm in its larger diameter in each inguinal location. It has to be accessible for administration after its localization using ultrasound scan.

Exclusion Criteria:

* Pregnant (positive to urine pregnancy test) or breastfeeding women.
* Subjects with history of any organic or psychic pathology in their records, physical exploration or any complementary test.
* Any relevant current pathology, including cancer, liver pathology, gastrointestinal dysfunction, renal alteration, respiratory pathology or active acute infectious problems.
* Chronic disorders or previous recurrent like hypertension, infections, cardiovascular, respiratory, endocrine, neurologic, hematologic, renal or liver disorders.
* Subjects treated four weeks before the first administration with any drug, medicinal plant or Consumer Health Care in a continue routine. It is not consider exclusion criteria a sporadic medication. The physician will study the interaction between the eASC with this medication.
* History of hypersensibility to drugs.
* Volunteers participants in other clinical trial within 4 months prior the start of the study.
* Blood or derivatives transfusion in 6 months before the trial.
* Known history of abuse of alcohol or other addictive substances(amount of alcohol allow as maximum in this trial is 0.5 liter of wine or two beers or amount in grams equivalent to this of any other alcoholic drink).
* Illegal drugs consumption during the month before the enrollment in the study or positive result to a drug test.
* Positive serology for B hepatitis virus (HbsAg), C hepatitis virus or HIV (Human Inmunodeficiency Virus).
* Subjects whose freedom depends on legal or administrative requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Local and systemic reaction to administration procedure | 29 days
  * Pain in administration area will be assessed by a visual analogical scale.
  * Medical exploration of the administration area will be performed to identify any skin reaction.
  * Inguinal scan will be performed to assess any lymphatic node modification.
  * Systemic tolerability will be measured by number of AE (Adverse Event) recorded at any time, including any alteration in laboratory parameters and/or physical exploration.

SECONDARY OUTCOMES:
Pharmacodynamic parameters | 29 days
  * Detection of reactive cells and antibodies against eASC
  * Lymphocyte subpopulations studies

CONTACTS AND LOCATIONS:
Overall Officials: Belén Sádaba, MD, Principal Investigator — Unidad de Investigación Clínica de la Clínica Universidad de Navarra
Locations (1):
- Unidad de Investigación Clínica de la Clínica Universidad de Navarra, Pamplona, Spain